CLINICAL TRIAL: NCT07093385
Title: The Effect of Intravitreal Faricimab in Patients With Refractory Macular Edema and Refractory Age Related Macular Degeneration
Brief Title: Intravitreal Faricimab in Patients With Refractory Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Duaa jabbar kadhim, principle investigator, University of Baghdad
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Ab2222
Record Dates: First submitted 2025-07-12; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — faricimab

STUDY DESIGN:
Intervention Model Description: All patients enrolled in this prospective study were a sample of Iraqi patients diagnosed with resistant AMD, DME or RVO edema. These patients diagnosed as primary non-responders to Bevacizumab, Lucentis or Aflibercept.Eligible participants received monthly intravitreal injections of Faricimab (6 mg/0.05 mL) for three months (loading dose) in a sterile environment, following standard aseptic protocols. Patients observation and examination repeated after One month from the last injection to assess treatment response (BCVA, IOP and SD-OCT re-evaluation).The response to Faricimab was determined using both anatomical (CRT) and functional (BCVA) markers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- faricimab (Experimental): Eligible participants received monthly intravitreal injections of Faricimab (6 mg/0.05 mL) for three months (loading dose) in a sterile environment, following standard aseptic protocols. Patients observation and examination repeated after One month from the last injection to assess treatment response (BCVA, IOP and SD-OCT re-evaluation).The response to Faricimab was determined using both anatomical (CRT) and functional (BCVA) markers
  Interventions: Drug: Faricimab Injection

INTERVENTIONS:
Drug: Faricimab Injection — Faricimab (6 mg/0.05 mL) for three months (loading dose) in a sterile environment,

SUMMARY:
This prospective study will include about 40 patients with resistant wet age-related macular degeneration (AMD), diabetic macular edema (DME), or retinal vein occlusion edema (RVO) edema.The inclusion criteria are that all patients must be 40 years old or older, diagnosed with active wet AMD or macular edema due to RVO or DME, and have received at least four previous monthly injections of anti-VEGF other than faricimab. All patients will be switched to receive four loading doses of intravitreal faricimab (6 mg) at 4-week intervals for four months. The response to faricimab will be assessed regarding visual acuity and central macular thickness.

DETAILED DESCRIPTION:
This prospective study will include about 40 patients with resistant wet age-related macular degeneration (AMD), diabetic macular edema (DME), or retinal vein occlusion edema (RVO) edema.

The inclusion criteria are that all patients must be 40 years old or older, diagnosed with active wet AMD or macular edema due to RVO or DME, and have received at least four previous monthly injections of anti-VEGF other than faricimab.

All patients will be switched to receive four loading doses of intravitreal faricimab (6 mg) at 4-week intervals for four months. The response to faricimab will be assessed regarding visual acuity (functionally), central macular thickness, and the presence of subretinal or intraretinal fluid (anatomically) by optical coherence tomography OCT and compared with pre-injection visual acuity and OCT.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 45 years or older 2. DME, RVO edema, or wet-AMD diagnosed by clinical evidence and optical coherence tomography angiography (OCTA).

  3. Previously treated with:
  * At least six doses of Avastin in DME or RVO edema cases or 3 dose of Avastin in AMD cases in the last year.
  * At least five doses of Eylea in DME or RVO edema cases or 3 dose of Eylea in AMD cases in the last year.

    4. Lack of significant anatomical or visual improvement (i.e., primary non-responders) 5. Willingness and ability to attend follow-up appointments and comply with treatment protocol.

Exclusion Criteria:

* 1. Inconsistent treatment history: missed a dose of anti-VEGF doses, or incomplete the three loading doses of Faricimab.

  2. Ocular comorbidities that could confound outcomes, such as:
  * Visually significant cataract as Grade 3+ or more.
  * Corneal opacity.
  * uveitis
  * Uncontrolled glaucoma (IOP > 25 mmHg on meds) with an increase in cup/disc ratio.
  * Other macular pathologies (e.g., macular hole, epiretinal membrane ERM) 3. Severe baseline vision loss (BCVA < 6/60).

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
central retinal thickness | one month after the last faricimab injection
  optical coherence tomography angiography

CONTACTS AND LOCATIONS:
Overall Officials: Duaa J Kadhim, Principal Investigator — University of Baghdad
Locations (1):
- Baghdad university, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code